CLINICAL TRIAL: NCT02854826
Title: Systems Addressing Frail Elders (SAFE) Care Implementation
Acronym: SAFE
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: UniHealth Foundation (Unknown); Ronald Reagan Medical Center (Unknown); Huntington Hospital (Other Government); Torrance Memorial (Unknown)
Responsible Party: Principal Investigator, Linda Burnes Bolton, DrPH, RN, FAAN, CNE, CNO, VP of Nursing, Cedars-Sinai Medical Center
Other Study IDs: 44067
Record Dates: First submitted 2016-07-22; First posted 2016-08-04 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2016-07

CONDITIONS: Frail Older Adutls
Keywords: Frail Older Adults, Interprofessional Team

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- UCLA Ronald Reagan Medical Center: Site 1 (UCLA Regan Medical Center): Leaders from nursing, pharmacy, social work/case management, physician, administration, performance improvement, information systems and the Nursing Research/Evidence Based Practice Council will implement, monitor and evaluate the SAFE Care model of care. Two nursing units will be identified for staff training in screening at-risk older adults. One units will be randomly selected to initiate the SAFE Care program. The "comparison" unit staff will screen for at-risk patients and continue usual high standard of care assessments and care planning. Both units will be closely followed with formative and summative evaluation data presented for local and all-site findings.
  Interventions: Other: SAFE Care model of care
- Huntington Hospital: Site 2 (Huntington Hospital): Leaders from nursing, pharmacy, social work/case management, physician, administration, performance improvement, information systems and the Nursing Research Council/ Evidence Based Practice will implement, monitor and evaluate the SAFE Care model of care. Two nursing units will be identified for staff training in screening at-risk older adults. One units will be randomly selected to initiate the SAFE Care program. The "comparison" unit staff will screen for at-risk patients and continue usual high standard of care assessments and care planning. Both units will be closely followed with formative and summative evaluation data presented for local and all-site findings.
  Interventions: Other: SAFE Care model of care
- Torrance Memorial Hospital: Site 3 (Torrance Memorial Hospital): Leaders from nursing, pharmacy, social work/case management, physician, administration, performance improvement, information systems and the Nursing Research/ Evidence Based Practice Council will implement, monitor and evaluate the SAFE Care model of care. Two nursing units will be identified for staff training in screening at-risk older adults. One units will be randomly selected to initiate the SAFE Care program. The "comparison" unit staff will screen for at-risk patients and continue usual high standard of care assessments and care planning. Both units will be closely followed with formative and summative evaluation data presented for local and all-site findings.
  Interventions: Other: SAFE Care model of care

INTERVENTIONS:
Other: SAFE Care model of care — SAFE Care Model Site Intervention:
  1. Endorse best practices for frail patients;
  2. Identify frail patients promptly using multi-dimensional screening and assessments;
  3. Employ interprofessional unit-based care team approach to frailty risk reduction during inpatient stay and create post-acute care transitions (PACT) plan recommendations;
  4. Develop electronic health record templates for patient-centered interprofessional frailty notes;
  5. Communicate PACT plans to primary care providers to promote safe transitions to the ambulatory setting and across the continuum of care.
  6. Increase awareness, improve management of frailty, and improve overall health and well-being for adults who are frail or at risk of becoming frail.

SUMMARY:
Systems Addressing Frail Elders (SAFE) Care is a nurse-led interprofessional team model to rapidly identify and provide safe and effective inpatient care to high risk older adults and help support their successful transition back to the community. Developed and demonstrated to be effective in one hospital - the model is now being disseminated and studied in three additional hospitals (multiple organizational case study).

DETAILED DESCRIPTION:
Three Magnet hospitals in Los Angeles County (Huntington Hospital, Torrance Memorial Medical Center and Ronald Reagan UCLA Health System) are collaborating on this demonstration and evaluation project (Multiple Case-Study Design). The project will engage interprofessional hospital leadership; provide training and coaching in implementation processes of the SAFE Care model; and track outcome of the SAFE Care model as implemented in the three collaborating site hospitals (three case studies). The investigators hope to contribute to the existing state of the science in dissemination and implementation of evidenced-based innovations. The collective data from the three sites (collected through interviews with hospital leadership and staff and with de-identified patient data on program implementation outcomes) will provide information about the effectiveness of the implementation process and support further dissemination.

ELIGIBILITY:
Inclusion criteria:

Organizational Leadership Nursing Unit Leadership/staff Adults aged 65 years

Exclusion criteria:

65 years and older that are on hospice protocols or dying/comfort care protocols.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This project does not have a set recruitment/enrollment goal. Process evaluation information will be collected by interview and observation of leadership and staff at three implementation sites. Quality Improvement (QI) outcome data will be collected involving elderly patients (> 65 years) admitted to two med-surg units at each of the three collaborating sites over designated time periods: One month prior to implementation and six month after intervention. QI data from each hospital will be de-identified and submitted to core research team for analysis of patient outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Implementation of SAFE Care model. Decreased Length of Stay | Up to 24 months
  The purpose of this project is to spread a successful model for rapidly identifying high risk vulnerable adults during an acute inpatient episode and intervening as an interprofessional team. An added purpose is to engage and promote involvement of participating hospitals' nursing research and evidence-based practice nurse experts in evaluating, adapting, and disseminating the SAFE Care model principles. We will evaluate if there is replication of the findings of the previous research (a cluster randomized controlled trial) conducted at Cedars-Sinai; that is, reduced LOS, reduced hospital complications (increased patient safety) and reduced use of ICU days. The evaluation plan for this project strongly supports collection and sharing of data on the process and outcomes of implementation of SAFE Care.
Implementation of SAFE Care model. Reduced use of ICU days | Up to 24 months
  he purpose of this project is to spread a successful model for rapidly identifying high risk vulnerable adults during an acute inpatient episode and intervening as an interprofessional team. An added purpose is to engage and promote involvement of participating hospitals' nursing research and evidence-based practice nurse experts in evaluating, adapting, and disseminating the SAFE Care model principles. We will evaluate if there is replication of the findings of the previous research (a cluster randomized controlled trial) conducted at Cedars-Sinai; that is, reduced LOS, reduced hospital complications (increased patient safety) and reduced use of ICU days. The evaluation plan for this project strongly supports collection and sharing of data on the process and outcomes of implementation of SAFE Care.
Implementation of SAFE Care model. Reduced hospital complications | Up to 24 months
  he purpose of this project is to spread a successful model for rapidly identifying high risk vulnerable adults during an acute inpatient episode and intervening as an interprofessional team. An added purpose is to engage and promote involvement of participating hospitals' nursing research and evidence-based practice nurse experts in evaluating, adapting, and disseminating the SAFE Care model principles. We will evaluate if there is replication of the findings of the previous research (a cluster randomized controlled trial) conducted at Cedars-Sinai; that is, reduced LOS, reduced hospital complications (increased patient safety) and reduced use of ICU days. The evaluation plan for this project strongly supports collection and sharing of data on the process and outcomes of implementation of SAFE Care.

CONTACTS AND LOCATIONS:
Overall Officials: Lianna Z Ansryan, MSN, Study Director — Cedars Sinai

IPD SHARING:
Plan to Share IPD: No